CLINICAL TRIAL: NCT06741475
Title: Optimizing Activity Performance of Stroke Patients Through Caregiver-Assisted Rehabilitation With Strategy Training: A Feasibility Study
Brief Title: Feasibility Study of Caregiver-Assist Strategy Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Feng-Hang Chang, Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: N202407030
Record Dates: First submitted 2024-12-14; First posted 2024-12-19 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: Stroke rehabilitation; Caregiver; Strategy training; Activity function
MeSH Terms: conditions — Stroke | interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: A researcher is responsible for the randomization process and the results are coded with predefined IDs that investigators and outcomes assessors are unaware of the meaning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caregiver-Assisted Strategy Training (Experimental): Trained therapists visit each participant once or twice weekly for 60 minutes per visit. In a total of 10 sessions over a maximum of 10 weeks, CaST program includes the following active ingredients: self-selected activity-based goals, dynamic performance analysis, global strategy ("Goal-PlanDo-Check"), massed practice, variable practice, increasing task difficulty, explicit and implicit feedback, guided discovery, action observation, and social interaction.
  Interventions: Behavioral: Caregiver-Assist Strategy Training
- Education (Sham Comparator): Participants receive a dose-matched stroke education with 10 visits by well-trained research staff through face-to-face talks.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Caregiver-Assist Strategy Training — CaST is a home-based rehabilitation that guides both stroke survivors and their caregivers to implement strategy training for addressing real-life limitations after stroke. During the intervention, the caregiver not only supervises the participant but also co-participates in the practice by instructing on when and how to be an assistant and facilitator when the stroke survivor executes their practice plan.
  Other Names: CaST
  Arms: Caregiver-Assisted Strategy Training
Behavioral: Education — Stroke-related information and knowledge that includes stroke subtypes and their etiology, risk factors of primary and secondary stroke, healthy lifestyles, common sequela, and adaptive skills for impaired functions are provided.
  Arms: Education

SUMMARY:
The goal of this study is to examine the feasibility of delivering an innovative intervention, caregiver-assisted strategy training (CaST), targeting enhancing activity functions in community-dwelling adults after stroke. The main questions it aims to answer are:

* Is CaST acceptable to stroke survivors with functional limitations?
* Does CaST show positive effects on functional outcomes?

Researchers will compare the CaST program to a control education program to investigate the interventional effect size for the selected stroke participants.

Participants will:

* Receive CAST or an education program 1 to 2 sessions per week until finishing 10 sessions.
* Be assessed clinical outcomes at 4 times: pre-intervention, post-intervention, 3-month, and 6-month follow-up.
* Be interviewed once after finishing their intervention.

DETAILED DESCRIPTION:
To address post-stroke activity limitations, intensive task-oriented rehabilitation is widely recommended across clinical guidelines. The caregiver is potentially able to play a facilitative role during the rehabilitation process. However, the best way to integrate caregivers into task-oriented rehabilitation is largely unknown. To address this gap, this preliminary study aims to assess the feasibility of a newly developed intervention, caregiver-assisted strategy training (CaST), in enhancing the activity performance of stroke survivors.

A mixed-methods (quantitative and qualitative) design, including a repeated measures design, is used in this feasibility study. A procedure of randomization with minimization will be conducted by a researcher who is independent of the investigation and outcome assessments. Eligible stroke survivors and their caregivers will be recruited from collaborative hospitals in Northern Taiwan and randomly assigned with even possibility. Longitudinal evaluations will be conducted at baseline (T1), post-intervention (T2), 3-month (T3), and 6-month (T4) follow-ups. Standardized assessments such as the Activity Measure for Post-Acute Care (AMPAC), the Participation Measure-3 Domains, 4 Dimensions (PM-3D4D), EuroQol-5D (EQ-5D), Stroke Self-Efficacy Questionnaires (SSEQ), Fugl-Meyer Assessment (FMA), Montreal Cognitive Assessment (MoCA), and Goal Attainment Scaling (GAS) will be used to assess outcomes at baseline, post-intervention, and 3-month and 6-month follow-ups. The feasibility indicators, such as recruitment rates and intervention attendance and adherence, will be evaluated by questionnaires, field notes, and qualitative interviews after the interventions are completed. Quantitative data will be analyzed using multiple linear regression models and mixed-effects regression models. Furthermore, qualitative in-depth interviews with participants, caregivers, and therapists will be conducted post-intervention. These interviews will explore experiences, satisfaction, and perceived effectiveness of the intervention. Transcribed data will undergo coding by two independent coders and subsequent analysis through the thematic analysis method.

ELIGIBILITY:
Inclusion Criteria:

* Being willing to provide informed consent
* Diagnosis with ischemic and/or hemorrhagic stroke
* Modified Rankin Scale (mRS) ranges from 2 to 4
* Rehabilitation frequency less than 3 days per week
* Having a healthy caregiver

Exclusion Criteria:

* Undergoing palliative care
* Major diseases or severe conditions influencing study participation, such as global aphasia, dementia, multiple organ failure, immobilization due to fracture, etc Moderate post-stroke cognitive impairment, with Montreal Cognitive Assessment score <22
* Pre-stroke mRS > 1
* Participating in other interventional study concurrently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Activity Measure for Post-Acute Care (AM-PAC) Outpatient Short Forms | 4 time points: baseline (T1), from baseline to the end of intervention at 5-10 weeks (T2), from the end of intervention to 3-month follow-up (T3), from the end of intervention to 6-month follow-up (T4)
  The AM-PAC measures the difficulty is performing three activity domains: Basic Mobility (18 activities), Daily Activity (15 activities), and Applied Cognition (19 activities) on a 4-point scale. In this trial, Applied Cognition domain is viewed as a secondary outcome. A trained research assistant performs AM-PAC face-to-face with participants. We determine the AM-PAC as the primary outcome due to its effect size from the between-group comparison will be used in developing the further efficacy trial.

SECONDARY OUTCOMES:
Participation Measure-3 Domains, 4 Dimensions (PM-3D4D) | 4 time points: baseline (T1), from baseline to the end of intervention at 5-10 weeks (T2), from the end of intervention to 3-month follow-up (T3), from the end of intervention to 6-month follow-up (T4)
  PM-3D4D consists of 24 items for evaluating three domains of participation, which are community, productivity, and social. Participants will be asked to rate all items on the four distinct dimensions: (1) diversity, (2) frequency, (3) desire for change, and (4) perceived difficulty. A trained research assistant performs PM-3D4D face-to-face with participants.
EuroQol-5D-3L (EQ-5D-3L) | 4 time points: baseline (T1), from baseline to the end of intervention at 5-10 weeks (T2), from the end of intervention to 3-month follow-up (T3), from the end of intervention to 6-month follow-up (T4)
  EuroQol-5D-3L (EQ-5D-3L) is a self-reported measurement that assesses participants' health-related quality of life across five domains: mobility, self-care, usual activity, pain/discomfort, anxiety/depression. In each domain, the assessment utilizes three levels to indicate the extent of problem: no problem, moderate problems, and extreme problems. A trained research assistant performs EQ-5D-3L face-to-face with participants.
Stroke Self-Efficacy Questionnaires (SSEQ) | 4 time points: baseline (T1), from baseline to the end of intervention at 5-10 weeks (T2), from the end of intervention to 3-month follow-up (T3), from the end of intervention to 6-month follow-up (T4)
  SSEQ measures individual confidence in functional performance after stroke [64]. It contains 13 items, and each item is rated on a 10-point scalar from 0 (not at all confident) to 10 (very confident). A trained research assistant performs SSEQ face-to-face with participants.
Fugl-Meyer Assessment (FMA) | 4 time points: baseline (T1), from baseline to the end of intervention at 5-10 weeks (T2), from the end of intervention to 3-month follow-up (T3), from the end of intervention to 6-month follow-up (T4)
  FMA measures the motor impairments of hemiplegia and includes a proximal subscale of upper extremity (0-42 points) for the shoulder/elbow/forearm, distal subscale of upper extremity (0-24 points) for the wrist/hand, and a lower extremity subscale (0-34 points) A trained research assistant performs FMA face-to-face with participants.
Montreal Cognitive Assessment (MoCA) | 4 time points: baseline (T1), from baseline to the end of intervention at 5-10 weeks (T2), from the end of intervention to 3-month follow-up (T3), from the end of intervention to 6-month follow-up (T4)
  MoCA with 30 items evaluates the cognitive functions. This assessment covers domains such as visuospatial/executive skills, naming, memory, attention, language, abstraction, delayed recall, and orientation. A trained research assistant performs MoCA face-to-face with participants.
Goal Attainment Scale | 4 time points: baseline (T1), from baseline to the end of intervention at 5-10 weeks (T2), from the end of intervention to 3-month follow-up (T3), from the end of intervention to 6-month follow-up (T4)
  GAS is used to quantify the achievement of goals. A trained research assistant performs GAS face-to-face with participants.
Client Satisfaction Questionnaire | At the end of intervention, 5 to 10 weeks from the baseline
  To quantify the participants' satisfaction about the intervention

OTHER OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | At baseline, within 4 weeks after enrollment
  NIHSS is used to indicate participants' stroke severity before intervention
Berg Balance Scale (BBS) | At baseline, within 4 weeks after enrollment
  BBS is used to indicate participants' balance function before intervention
Hospital Anxiety and Depression Scale (HADS) | At baseline, within 4 weeks after enrollment
  HADS is used to indicate participants' mood status before intervention
modified Rankin Scale (mRS) | 4 time points: baseline (T1), from baseline to the end of intervention at 5-10 weeks (T2), from the end of intervention to 3-month follow-up (T3), from the end of intervention to 6-month follow-up (T4)
  mRS is used to indicate participants' global disability

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Heng Chang, ScD, Principal Investigator — Graduate Institute of Injury Prevention and Control, Taipei Medical University
Locations (3):
- Taiwan (3):
  - Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, New Taipei City
  - Taipei Medical University Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No